CLINICAL TRIAL: NCT03615664
Title: The Efficacy of Bendamustine, Gemcytabine, Dexamethasone (BGD) Salvage Chemotherapy With autoSCT Consolidation in Advanced Classical HL Patients Not Responding to ABVD - Multicentre Phase II Clinical Study - PLRG-HL1
Brief Title: The Efficacy of Salvage BGD With autoSCT Consolidation in Advanced Classical HL Patients Not Responding to ABVD
Acronym: BURGUND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Polish Lymphoma Research Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLRG-HL1
Record Dates: First submitted 2018-07-19; First posted 2018-08-06 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Hodgkin's Lymphoma
Keywords: Lymphoma; Immunochemotherapy; Salvage therapy; Bendamustine; Gemcitabine; Dexamethasone; Hodgkin's Lymphoma; ASCT
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Bendamustine Hydrochloride; Gemcitabine; Dexamethasone; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BGD therapy (Experimental): Bendamustine, Gemcitabine, Dexamethasone
  Interventions: Drug: Bendamustine; Drug: Gemcitabine; Drug: Dexamethasone; Diagnostic Test: PET/CT; Procedure: Autologous Stem Cell Transplant

INTERVENTIONS:
Drug: Bendamustine — Bendamustine (B) 90 mg/m2 i.v. day 1, 2
  Other Names: Treanda
Drug: Gemcitabine — Gemcitabine (G) 800 mg/m2 i.v. day 1, 4
  Other Names: Gemzar
Drug: Dexamethasone — Dexamethasone (D) 40 mg i.v./p.o. day 1,2,3,4
Diagnostic Test: PET/CT — PET scan/CT must be performed after first 2 courses of BGD treatment. Results evaluation:
  * in case of a CMR/CR or PMR/PR, ASCT must be performed within 3 months after the end of BGD treatment
  * in case of SMD - exclusion from the trial
  * in case of PMD - exclusion from the trial
Procedure: Autologous Stem Cell Transplant — Must be performed within 3 months after the end of BGD treatment.
  When it is not possible to perform ASCT, despite CMR or PMR response, within 3 months after second course of BGD treatment, it is permissible to extend the therapy up to 4 cycles. PET scan/CT must be repeated before performing ASCT.
  Other Names: ASCT

SUMMARY:
The objective of the study is evaluation of efficacy of Bendamustine, Gemcytabine, Dexamethasone (BGD) salvage therapy with autologus stem cell transplantation (ASCT) consolidation in advanced classical Hodgkin lymphoma patients not responding to ABVD therapy.

DETAILED DESCRIPTION:
Treatment regimen:

Bendamustine (B) 90 mg/m2 iv day 1, 2 Gemcytabine (G) 800 mg/m2 iv day 1, 4 Dexamethasone (D) 40 mg iv/po day 1,2,3,4

Course of treatment every 21-28 days, 4 courses of treatment max; next round of treatment may be given if ANC>1000/μl and PLT>75000/μl. Up to 7-day delay is permitted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Classical Hodgkin's Lymphoma treated with ABVD regimen with PET scan/CT performed before, during and after treatment, and also one of the following:

  * positive result (Deauville 4 and 5) of early PET scan after 2 ABVD courses
  * disease progression or relapse after first-line ABVD treatment or ABVD and radiotherapy combination treatment
* No contraindications for salvage chemotherapy and ASCT
* At least one measurable malignancy
* ECOG performance status ≤ 3
* Written signed and dated informed consent prior to any study procedures being performed

Exclusion Criteria:

* Non-Classical Hodgkin's Lymphoma
* Other than ABVD first-line treatment, preceding patient's inclusion
* Lack of PET scans performed in accordance with inclusin criteria during ABVD treatment
* Transformation of Hodgkin's Lymphoma
* Central Nervous System (CNS) Metastases
* Contraindications for ASCT or lack of patient's consens for the procedure
* Second malignancy - active or cured less than 5 years prior
* Uncontrolled diabetes
* Hepatic impairment (bilirubin concentration ≥ 1.5 x ULN, SGOT > 5 x ULN), if non-realted to the lymphoma or Gilbert's syndrome
* HIV infection
* Active HBV or HCV infection. Subjects who have had Hepatitis B and are abHBC positive, need to undergo HBV DNA test using a Polymerase Chain Reaction (PCR) technique and be applied appropriate preventive treatment.
* Pregnancy or lactation
* Hypersensitivity to any of the drugs
* Lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
ORR (overall response rate) | Evaluated at the end of Cycle 2 of BGD (every cycle is 21-28 days)
  CR (complete response) + PR (partial response)
PFS (progression-free survival) | Time measured from date of of Cycle 2 of BGD treatment (every cycle is 21-28 days) until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Staying free of disease progression.

SECONDARY OUTCOMES:
OS (overall survival) | Time measured from Day 1 of Cycle 1 of BGD treatment (every cycle is 21-28 days) until the date of death from any cause, assessed up to 24 months (measured for patients that have undergone ASCT after BGD tratment).
  The length of time from the start of treatment, that patients diagnosed with the disease are still alive.
OMRR (overall metabolic response rate) | Evaluated a the end of Cycle 2 of BGD treatment (every cycle is 21-28 days) and after ASCT (up to 150 days after Day 1 of Cycle 1 of BGD treatment).
  OMRR= CMR (complete metabolic response) + PMR (partial metabolic response)
BGD tolerability assessment. | 24 months from the start of BGD treatment
  Number of participants with treatment-related adverse events and serious adverse events.
MR (mobilization rate) | Evaluated after the end of Cycle 2 of BGD (every cycle is 21-28 days), before tranplantation (up to Day 150 of treatment).
  Evaluation of stem cells mobilization efficacy in patients on BGD regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Giebel, Prof., Study Director — PLRG's Chairman
Locations (13):
- Poland (13):
  - Oddział Kliniczny Onkologii, Centrum Onkologii im. Prof. F. Łukaszczyka, Bydgoszcz
  - Klinika Hematologii i Transplantologii, Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Centrum Onkologii - Instytut im. M. Skłodowskiej-Curie, Oddział w Gliwicach, Gliwice
  - Oddział Chorób Wewnętrznych i Chemioterapii Onkologicznej, Samodzielny Publiczny Szpital Kliniczny im. A.Mielęckiego, Katowice
  - Oddział Hematologii, Szpital Specjalistyczny im. Rydygiera, Krakow
  - Klinika Hematoonkologii i Transplantacji Szpiku, Samodzielny Publiczny Szpital Kliniczny nr 1, Lublin
  - Oddział Hematologii, Samodzielny Publiczny ZOZ MSWiA z Warmińsko-Mazurskim Centrum Onkologii, Olsztyn
  - Oddział Hematologii i Onkologii Hematologicznej, Szpital Wojewódzki w Opolu, Opole
  - NU-MED Centrum Diagnostyki i Terapii Onkologicznej, Tomaszów Mazowiecki
  - Centrum Onkologii-Instytut im. M. Skłodowskiej-Curie, Warsaw
  - Klinika Chorób Wewnętrznych i Hematologii, Wojskowy Instytut Medyczny, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1, Wroclaw

IPD SHARING:
Plan to Share IPD: No